CLINICAL TRIAL: NCT03413683
Title: Frailty in Older HIV-infected Individuals in Hong Kong: Risk Factors and Association With Quality of Life and Mortality
Brief Title: Frailty in Older HIV-infected Individuals
Status: Recruiting | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Grace Lui, Clinical Assistant Professor, Chinese University of Hong Kong
Other Study IDs: Geri_HIV protocol v1 03Nov2017
Record Dates: First submitted 2018-01-23; First posted 2018-01-29 (Actual); Last update posted 2023-08-30 (Actual); Status verified 2023-08

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Peripheral blood samples
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Frailty has been proposed as a measure of biological (as opposed to chronological) aging. In this study the investigators plan to: (1) measure frailty in a cohort of older HIV-infected individuals in Hong Kong, and its association with mortality and quality of life; (2) identify risk factors predictive of development of frailty in HIV-infected individuals in Hong Kong; and (3) determine the outcomes of HIV-infected individuals in Hong Kong with and without frailty.

The following assessment will be done:

1. Physical examination including measuring height, weight, hip and waist circumference.
2. Grip strength, chair stand test, gait speed test, balance tests, and neurocognitive tests
3. Geriatric syndromes, screening for depression, disability and quality of life.
4. Blood tests during fasting state to measure metabolic parameters.

This is a prospective longitudinal observational study that lasts for 10 years.

ELIGIBILITY:
Inclusion Criteria:

* HIV infection with positive anti-HIV antibody
* Age ≥50 years

Exclusion Criteria:

* Refuses to consent

Min Age: 50 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: HIV-positive patients who attend Infectious Diseases clinic at Prince of Wales Hospital
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2018-04-01 (Actual); Primary Completion 2028-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Frailty | 10 years
  Frailty defined by frailty phenotype measurement, according to Fried (Fried et al., 2011) definition.

CONTACTS AND LOCATIONS:
Overall Officials: Grace Lui, Principal Investigator — CUHK
Locations (1):
- Prince of Wales Hospital, Shatin, Hong Kong

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Fried LP, Tangen CM, Walston J, Newman AB, Hirsch C, Gottdiener J, Seeman T, Tracy R, Kop WJ, Burke G, McBurnie MA; Cardiovascular Health Study Collaborative Research Group. Frailty in older adults: evidence for a phenotype. J Gerontol A Biol Sci Med Sci. 2001 Mar;56(3):M146-56. doi: 10.1093/gerona/56.3.m146. PMID 11253156